CLINICAL TRIAL: NCT07367113
Title: Effect of Peripheral Perfusion Index-guided Fluid Resuscitation on the Prevention of Acute Skin Failure in Elderly Critically Ill Patients: A Prospective, Randomized, Controlled Trial
Brief Title: Peripheral Perfusion Index-guided Fluid Resuscitation for Preventing Acute Skin Failure in Elderly Critically Ill Patients
Acronym: PPI-PROTECT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ying Wang (Other)
Collaborators: Affiliated Haian People's Hospital of Nantong University (Unknown)
Responsible Party: Sponsor-Investigator, Ying Wang, Clinical Professor, Nantong First People's Hospital
Organization: Nantong First People's Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: HAYY - 2025 - LW - 045
Record Dates: First submitted 2026-01-16; First posted 2026-01-26 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2026-01

CONDITIONS: Sepsis; Septic Shock; Acute Skin Failure
MeSH Terms: conditions — Sepsis; Shock, Septic

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- eripheral Perfusion Index-guided Fluid Resuscitation Protocol (Experimental)
  Interventions: Other: Peripheral Perfusion Index-guided Fluid Resuscitation Protocol
- Conventional Fluid Resuscitation Group (Active Comparator)
  Interventions: Other: Conventional Goal-Directed Fluid Resuscitation

INTERVENTIONS:
Other: Peripheral Perfusion Index-guided Fluid Resuscitation Protocol — In addition to achieving conventional macro-hemodynamic goals (mean arterial pressure ≥65 mmHg, etc.), a resuscitation protocol targeting a Peripheral Perfusion Index (PPI) value ≥1.4 is implemented. PPI is continuously monitored via a finger pulse oximeter. If PPI remains below 1.4 for >30 minutes, a fluid responsiveness assessment (e.g., passive leg raising test) is performed. Fluid boluses (balanced crystalloid) are administered only if the patient is fluid-responsive. Otherwise, vasoactive agents are optimized.
  Arms: eripheral Perfusion Index-guided Fluid Resuscitation Protocol
Other: Conventional Goal-Directed Fluid Resuscitation — Fluid resuscitation is performed according to the Surviving Sepsis Campaign International Guidelines. Resuscitation targets include: mean arterial pressure ≥65 mmHg, central venous pressure 8-12 mmHg, urine output ≥0.5 mL·kg-¹·h-¹, and normalization/decreasing trend of serum lactate. The type, rate, and volume of fluid administration are determined by the treating physician based on these standard macro-hemodynamic and perfusion parameters.
  Arms: Conventional Fluid Resuscitation Group

SUMMARY:
This prospective, randomized, controlled trial aimed to evaluate whether fluid resuscitation guided by the Peripheral Perfusion Index (PPI) could reduce the incidence of Acute Skin Failure (ASF) in elderly critically ill patients. A total of 216 patients aged ≥65 years with sepsis or other types of shock requiring early aggressive fluid resuscitation were enrolled and randomly assigned in a 1:1 ratio to either the PPI-guided resuscitation group or the conventional resuscitation group. The intervention group targeted maintaining PPI ≥1.4 in addition to conventional hemodynamic goals, while the control group followed standard resuscitation protocols. The primary outcome was the incidence of ASF within 7 days of ICU admission, diagnosed according to NPUAP/EPUAP (2014) criteria. Secondary outcomes included time to ASF occurrence, lactate clearance, cumulative fluid balance, organ function, and long-term prognosis.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 65 years.
2. Diagnosis of sepsis (according to Sepsis-3 criteria) or other types of shock requiring early and aggressive fluid resuscitation.
3. APACHE II score ≥ 15 at ICU admission.
4. Expected ICU length of stay ≥ 72 hours.
5. Written informed consent obtained from the patient or their legally authorized representative.

Exclusion Criteria:

1. Pre-existing stage III or higher pressure injury or skin necrosis at the time of enrollment.
2. Severe dermatological disease or peripheral vascular disease that could interfere with the assessment of skin or peripheral perfusion.
3. Inability to perform continuous finger pulse oximetry monitoring (e.g., due to bilateral finger injury, amputation, or severe peripheral edema).
4. Contraindications to liberal fluid resuscitation (e.g., acute cardiogenic pulmonary edema, severe heart failure with fluid overload).
5. Expected survival < 24 hours due to terminal illness or irreversible condition. Concurrent participation in another interventional clinical trial.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 216 (Estimated)
Dates: Start 2025-01-01 (Actual); Primary Completion 2026-02 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Incidence of Acute Skin Failure | From ICU admission up to 7 days
  Proportion of patients who develop new-onset Acute Skin Failure (ASF) within 7 days after ICU admission. ASF is diagnosed and staged according to the NPUAP/EPUAP (2014) criteria.

SECONDARY OUTCOMES:
Time to Acute Skin Failure (ASF) Onset | From ICU admission up to 7 days
  Number of days from ICU admission to the first diagnosis of ASF (assessed in patients who develop ASF)
Maximum Stage of Acute Skin Failure | From ICU admission up to 7 days
  The most severe stage of ASF (according to NPUAP/EPUAP 2014 criteria) observed within 7 days after ICU admission
Lactate Clearance Rate at 6 Hours | Baseline and 6 hours after resuscitation initiation
  Percentage decrease in serum lactate concentration from baseline to 6 hours after initiation of resuscitation
Lactate Clearance Rate at 24 Hours | Baseline and 24 hours after resuscitation initiation
  Percentage decrease in serum lactate concentration from baseline to 24 hours after initiation of resuscitation
Cumulative Fluid Balance at 72 Hours | From ICU admission up to 72 hours
  Net fluid balance (total fluid intake minus total output) calculated over the first 72 hours of ICU stay
Incidence of Acute Kidney Injury | From ICU admission up to 7 days
  Proportion of patients who develop AKI according to KDIGO criteria within 7 days after ICU admission
Duration of Mechanical Ventilation | From ICU admission until ICU discharge, up to 90 days
  Total number of days requiring invasive mechanical ventilation during ICU stay
Length of ICU Stay | From ICU admission until ICU discharge, up to 90 days
  Total number of days from ICU admission to ICU discharge
28-Day All-Cause Mortality | From ICU admission up to 28 days
  Proportion of patients who die from any cause within 28 days after ICU admission
90-Day All-Cause Mortality | From ICU admission up to 90 days
  Proportion of patients who die from any cause within 90 days after ICU admission
Barthel Index at Hospital Discharge | At hospital discharge, up to 90 days after ICU admission
  Score of the Barthel Index (a measure of activities of daily living) assessed at the time of hospital discharge in surviving patients. Range: 0-100, higher scores indicate greater independence
Total Hospitalization Costs | From hospital admission to hospital discharge, up to 90 days
  Total direct medical costs incurred during the index hospitalization, expressed in local currency
30-Day Unplanned Readmission Rate | 30 days after hospital discharge
  Proportion of patients who have an unplanned readmission to any hospital within 30 days after hospital discharge
Incidence of Resuscitation-Related Serious Adverse Events | From ICU admission until ICU discharge, up to 90 days
  Proportion of patients who experience serious adverse events related to fluid resuscitation (e.g., new-onset cardiogenic pulmonary edema, arrhythmia requiring intervention) during the ICU stay

CONTACTS AND LOCATIONS:
Locations (1):
- Nantong First People's Hospital, Nantong, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No
We may have further research, and we may not consider releasing the research data until the results are announced